CLINICAL TRIAL: NCT00382161
Title: Influence of Treatment With the HMG-CoA-Reductase Inhibitor Fluvastatin on Erectile Function in Patients With Cardiovascular Risk-Factors and Erectile Dysfunction
Brief Title: Improvement of Erectile Dysfunction by Fluvastatin in Patients With Cardiovascular Risk Factors
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: not enough patients meeting inclusion criteria
Sponsor: University Hospital, Saarland (Other)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 48/05; EudraCT-No.:2006-000284-28
Record Dates: First submitted 2006-09-27; First posted 2006-09-28 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Impotence
Keywords: impotence; erectile dysfunction; cardiovascular risk factor; statin
MeSH Terms: conditions — Erectile Dysfunction | interventions — Fluvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fluvastatin-sodium

SUMMARY:
The purpose of the study is to determine the effect of fluvastatin on penile arterial blood flow and erectile function in patients with arteriogenic ED and cardiovascular risk factors.

DETAILED DESCRIPTION:
Physiology of erection is mainly dependent on endothelial NO-production with consecutive activation of guanylate-cyclase. Pleiotropic effects of statins are well known regarding the increase of endothelial function. Thus, activation of endothelial NO-synthase could raise the activation of guanylate-cyclase with a consecutive relaxation of smooth muscle cells in the penile arteries and the corpus cavernosum leading to an improvement of erectile function. Therefore, statins are supposed to be effective in the treatment of erectile dysfunction, especially in patients with cardiovascular risk-factors with underlying endothelial dysfunction.

The effect of fluvastatin on penile blood-flow and erectile function in patients with arteriogenic erectile dysfunction and cardiovascular risk factors will be determined in a cross-over design. Patients were either treated with fluvastatin-sodium 80mg or placebo for 8 weeks. After a wash-out of 4 weeks, treatment will be switched (placebo / fluvastatin-sodium). Penile blood flow measurement and assessment of erectile function with the IIEF-5-score and the KEED-score will be performed at baseline, after 8 weeks of treatment, after 4 weeks wash-out and after cross-over treatment (8 weeks).

ELIGIBILITY:
Inclusion Criteria:

* male
* age > 18 years
* arteriogenic erectile dysfunction (penile blood flow - peak systolic velocity<30cm/s, diastolic velocity<5cm/s)
* two or more cardiovascular risk factors (smoking, hypertension, hyperlipoproteinaemia, family history of atherosclerosis, oral treated diabetes mellitus with a HbA1c<7%)
* stable course of disease without expected changes in medical treatment during the next 3 months
* written informed consent
* no statin-treatment so far

Exclusion Criteria:

* known hypersensitivity or anaphylaxis against a statin
* active liver disease or unclear increase of transaminases, cholestasis or myopathy
* acute cardiovascular event (myocardial infarction, stroke, PTCA, vascular surgery) within 3 months before randomization
* clinical signs of heart failure or reduced left ventricular function
* current treatment with lipid lowering drugs
* insulin dependent diabetes mellitus or orally treated diabetes mellitus with a HbA1c-value >6.9%
* erectile dysfunction due to hormone disorders
* known malignant tumor
* known disposition to priapism
* patients with morphological changes of the penis (i.e. deviation) or penis-prosthesis
* current treatment with anticoagulants
* current treatment with immunosuppressive drugs, phenytoin, erythromycin, gemfibrozil or nicotinic acid derivates
* absence or inability of written informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-10; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Penile blood flow (peak systolic velocity, resistance index, pulsatility index) after 8 weeks of treatment.

SECONDARY OUTCOMES:
Erectile function assessed with the IIEF-5 score (international index of erectile function) after 8 weeks of treatment.
Erectile function assessed with the KEED score (cologne questionnaire of erectile function) after 8 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Baumhäkel, MD, Principal Investigator — University Hospital of the Saarland; Michael Böhm, MD, Principal Investigator — University Hospital of the Saarland; Martin Gerber, MD, Principal Investigator — University Hospital of the Saarland; Michael Stöckle, MD, Principal Investigator — University Hospital of the Saarland
Locations (1):
- University Hospital of the Saarland, Homburg, Saarland, Germany

REFERENCES:
- [Background] Diagnosis and treatment of early melanoma. NIH Consensus Development Conference. January 27-29, 1992. Consens Statement. 1992 Jan 27-29;10(1):1-25. PMID 1515516
- [Background] Kinsey AC, Pomeroy WR, Martin CE. Sexual behavior in the human male. 1948. Am J Public Health. 2003 Jun;93(6):894-8. doi: 10.2105/ajph.93.6.894. No abstract available. PMID 12773346
- [Background] Virag R, Bouilly P, Frydman D. Is impotence an arterial disorder? A study of arterial risk factors in 440 impotent men. Lancet. 1985 Jan 26;1(8422):181-4. doi: 10.1016/s0140-6736(85)92023-9. PMID 2857264
- [Background] Feldman HA, Goldstein I, Hatzichristou DG, Krane RJ, McKinlay JB. Impotence and its medical and psychosocial correlates: results of the Massachusetts Male Aging Study. J Urol. 1994 Jan;151(1):54-61. doi: 10.1016/s0022-5347(17)34871-1. PMID 8254833
- [Background] Braun M, Wassmer G, Klotz T, Reifenrath B, Mathers M, Engelmann U. Epidemiology of erectile dysfunction: results of the 'Cologne Male Survey'. Int J Impot Res. 2000 Dec;12(6):305-11. doi: 10.1038/sj.ijir.3900622. PMID 11416833
- [Background] Grimm RH Jr, Grandits GA, Prineas RJ, McDonald RH, Lewis CE, Flack JM, Yunis C, Svendsen K, Liebson PR, Elmer PJ. Long-term effects on sexual function of five antihypertensive drugs and nutritional hygienic treatment in hypertensive men and women. Treatment of Mild Hypertension Study (TOMHS). Hypertension. 1997 Jan;29(1 Pt 1):8-14. doi: 10.1161/01.hyp.29.1.8. PMID 9039073
- [Background] Wei M, Macera CA, Davis DR, Hornung CA, Nankin HR, Blair SN. Total cholesterol and high density lipoprotein cholesterol as important predictors of erectile dysfunction. Am J Epidemiol. 1994 Nov 15;140(10):930-7. doi: 10.1093/oxfordjournals.aje.a117181. PMID 7977280
- [Background] Chitaley K, Wingard CJ, Clinton Webb R, Branam H, Stopper VS, Lewis RW, Mills TM. Antagonism of Rho-kinase stimulates rat penile erection via a nitric oxide-independent pathway. Nat Med. 2001 Jan;7(1):119-22. doi: 10.1038/83258. PMID 11135626
- [Background] Buyukafsar K, Un I. Effects of the Rho-kinase inhibitors, Y-27632 and fasudil, on the corpus cavernosum from diabetic mice. Eur J Pharmacol. 2003 Jul 11;472(3):235-8. doi: 10.1016/s0014-2999(03)01905-8. PMID 12871759
- [Background] Wassmann S, Ribaudo N, Faul A, Laufs U, Bohm M, Nickenig G. Effect of atorvastatin 80 mg on endothelial cell function (forearm blood flow) in patients with pretreatment serum low-density lipoprotein cholesterol levels <130 mg/dl. Am J Cardiol. 2004 Jan 1;93(1):84-8. doi: 10.1016/j.amjcard.2003.09.018. PMID 14697473
- [Background] Nangle MR, Cotter MA, Cameron NE. Effects of rosuvastatin on nitric oxide-dependent function in aorta and corpus cavernosum of diabetic mice: relationship to cholesterol biosynthesis pathway inhibition and lipid lowering. Diabetes. 2003 Sep;52(9):2396-402. doi: 10.2337/diabetes.52.9.2396. PMID 12941781
- [Background] Rosen RC, Cappelleri JC, Smith MD, Lipsky J, Pena BM. Development and evaluation of an abridged, 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool for erectile dysfunction. Int J Impot Res. 1999 Dec;11(6):319-26. doi: 10.1038/sj.ijir.3900472. PMID 10637462
- [Background] Speel TG, van Langen H, Wijkstra H, Meuleman EJ. Penile duplex pharmaco-ultrasonography revisited: revalidation of the parameters of the cavernous arterial response. J Urol. 2003 Jan;169(1):216-20. doi: 10.1016/S0022-5347(05)64071-2. PMID 12478139
- [Background] Aversa A, Isidori AM, Spera G, Lenzi A, Fabbri A. Androgens improve cavernous vasodilation and response to sildenafil in patients with erectile dysfunction. Clin Endocrinol (Oxf). 2003 May;58(5):632-8. doi: 10.1046/j.1365-2265.2003.01764.x. PMID 12699447
- [Background] Laufs U, Wassmann S, Hilgers S, Ribaudo N, Bohm M, Nickenig G. Rapid effects on vascular function after initiation and withdrawal of atorvastatin in healthy, normocholesterolemic men. Am J Cardiol. 2001 Dec 1;88(11):1306-7. doi: 10.1016/s0002-9149(01)02095-1. No abstract available. PMID 11728362